CLINICAL TRIAL: NCT06356038
Title: Phrenic Nerve Infiltration: a Good Practice to Combine Pulmonary Expansion and Pain Control in Patients With High-risk of Prolonged Air Leak
Brief Title: Phrenic Nerve Infiltration: Pulmonary Expansion and Pain Control
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera "Sant'Andrea" (Other)
Responsible Party: Principal Investigator, Beatrice Trabalza Marinucci, MD, Principal Investigator, Azienda Ospedaliera "Sant'Andrea"
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prot. n. 76 SA/2022
Record Dates: First submitted 2024-03-22; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Prolonged Air Leak; Post-operative Pain
Keywords: prolonged air leak; phrenic nerve; local anaesthetic
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (phrenic nerve infiltration) (Experimental): Patients received intra-operative phrenic nerve infiltration with local anesthetic
  Interventions: Procedure: intra-operative phrenic nerve infiltration
- Group B (no phrenic nerve infiltration) (No Intervention): Patients did not receive intra-operative infiltration

INTERVENTIONS:
Procedure: intra-operative phrenic nerve infiltration — patients received the intra-operative infiltration of phrenic nerve by the surgeon who injected 10 ml of Ropivacaine 0.75% (the same procedure routinely adopted in our clinical practice for local analgesia at the level of the intercostal space) in the peri-neurotic pericardial fat, near the diaphragm. Infiltration is made with a deflated lung, after pulmonary resection and chest tube insertion.
  Arms: Group A (phrenic nerve infiltration)

SUMMARY:
Between January 2021-2023, 65 consecutive patients at risk for PAL (defined in accordance to "2019 Society of Thoracic Surgery score-criteria of PAL") underwent lung resection (lobectomy or sublobar resection) for malignancy. 5 patients were lost. The remaining have been assigned with a 1:2 randomization into: group A (22 patients), received intra-operative phrenic nerve infiltration with Ropivacaine 10 mg/ml in the peri-neurotic fat on the pericardium and group B (38 patients), did not receive infiltration. Data on hemidiaphragm elevation, air leaks, pain at 24 and 72 hours post-surgery, shoulder pain, length of hospital stay, length of chest tube permanence, were retrospectively collected and compared.The aim of the study is to investigate the effect of intra-operative phrenic nerve infiltration with long acting anesthetic in patients at high risk for PAL, improving pulmonary expansion after surgery, and reducing air leaks, while controlling post-operative pain.

DETAILED DESCRIPTION:
This prospective randomized trial received approbation by the institutional review board (Prot. n. 76 SA/2022 RIF. CE 6682/2022) and was conducted in accordance with the Declaration of Helsinki. Written informed consent was obtained from all patients.

Patients were defined at risk for PAL in accordance with "2019 Society of Thoracic Surgery score-criteria of PAL". This is an aggregate score specifically designed for lung resection, assigning an odd risk to each patient based on the most common predictors for prolonged air leak including: Body Mass Index <_25.5 kg/m2 (7 points); lobectomy or bilobectomy (6 points); forced expiratory volume in 1 second (FEV1) </= 70% (5 points); male sex (4 points); right upper lobe (3 points). A total score > 17 is considered high risk for PAL.

All patients received pre-operative physical examination, routine blood tests, pulmonary functional test (spirometry and arterial blood gas analysis) and cardiac tests according to the personal clinical history. Imaging collection includes Total Body Computed Tomography (CT) and Positron Emission Tomography (PET). Central tumours required bronchoscopy to assess an eventual endobronchial invasion and to obtain histological diagnosis. If N1/N2 staging was clinically suspected, patients underwent Endo-Bronchial Ultra-Sonography (EBUS) with eventual Trans-Bronchial Needle Aspiration (TBNA) or mediastinoscopy.

Exclusion criteria for the study were: wedge resections, pneumonectomy, neoplasms infiltrating diaphragm and/or chest wall, patients with congenital or acquired neurological diseases, chronic pain, osteo-muscular pathologies affecting the shoulder.

All candidate patients for surgery underwent lung resection with a muscle sparing thoracotomy (lateral 5-6 cm incision on the fifth intercostal space), to reduce bias due by different surgical approaches on the post-operative pain.

In group A, patients received the intra-operative infiltration of phrenic nerve by the surgeon who injected 10 ml of Ropivacaine 0.75% (the same procedure routinely adopted in our clinical practice of local analgesia at the level of intercostal spaces) in the peri-neurotic pericardial fat, near the diaphragm. Infiltration is made with a deflated lung, after pulmonary resection and chest tube insertion.

Chest tubes were connected to a pleur-evac device with a system to register air leaks (DrentechTM Palm Evo, Redax).

All patients received Chest X-Rays in post-operative day 1, 3, 5. Pain control was assessed using Numeric Rating Scale (NRS), from 0 (no pain) to 10 (maximum level of pain) at 24-hors and 72-hours from surgery. Even the need for additional antalgic medicaments was registered. All patients started pulmonary rehabilitation programs (mobilization and respiratory exercises) on post-operative day 1.

Data were collected and stored in an Excel database (Microsoft Corp, Redmond, Wash) and were analyzed using statistical package SPSS, version 25.0 (SPSS Software, IBM Corp., Armonk, NY, USA). Data collected were then analyzed and compared between the two groups. Values were expressed as mean ± standard deviation (SD) for continuous variables and as absolute number and percentage in categorical variables. Comparison of categorical variables was performed by c2 test using Fischer exact test. Comparison of qualitative variables was performed by student t-test. Significance was defined as a P value of less than 0.05. The adjusted odd ratios (ORs) and 95% confidence intervals (CI) were calculated to estimate and measure the association using 1000 bootstrapping samples.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by lung cancer eligible for surgery
* patients with high risk for post-operative prolonged air leaks: Body Mass Index <_25.5 kg/m2 (7 points); lobectomy or bilobectomy (6 points); forced expiratory volume in 1 second (FEV1) </= 70% (5 points); male sex (4 points); right upper lobe (3 points). A total score > 17 is considered high risk for PAL

Exclusion Criteria:

* metastatic desease
* patients not eligible for surgery because low performance status
* pneumonectomy/ wedge resections
* tumors infiltrating phrenic nerve/ diaphragm
* patients with neurological disorders causing chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2025-01-02 (Estimated); Study Completion 2025-01-02 (Estimated)

PRIMARY OUTCOMES:
rate of pulmonary expansion due by phrenic nerve intra-operative local anaesthetic infiltration | two years
  Rate of pulmonary re-expansion that was defined complete or near complete if lung achieved the 90% of lung surface to the XR; incomplete if lung surface was inferior to 90%. The rate of lung surface is calculated evaluating the "mean interpleural distance": the measurement corresponds to the average of the distances between lung and chest wall calculated at three points (apex, costophrenic sinus, midpoint) in a chest XR; from the average of the three measurements, the rate of lung collapse and the rate of expansion are estimated.

SECONDARY OUTCOMES:
rate of post-operative pain control after intra-operative phrenic nerve infiltration with local anaesthetic | two years
  Pain control was assessed using Numeric Rating Scale (NRS), from 0 (no pain) to 10 (maximum level of pain) at 24-hors and 72-hours from surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera "Sant'Andrea", Roma, Italy

IPD SHARING:
Plan to Share IPD: No